CLINICAL TRIAL: NCT07034235
Title: Clinical Evaluation of the Effect of Wet and Overwet Dentin Using Two Universal Adhesives in Restorations of Non-carious Cervical Lesions: Double Blind Randomized Clinical Trial
Brief Title: Effect of Wet and Overwet Dentin on the Clinical Performance of Two Universal Adhesive Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Principal Investigator, Mario Felipe Gutiérrez Reyes, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F142025
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Non-carious Cervical Lesions
Keywords: Dental bonding; Tooth erosion; Tooth Wear; Adhesive systems; Dentinal moisture
MeSH Terms: conditions — Tooth Erosion; Tooth Wear

STUDY DESIGN:
Intervention Model Description: This is a four-arm, double-blind, randomized controlled clinical trial. Control group 1: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Ambar Universal APS Plus; FGM) on wet dentin in the etch-and-rinse application strategy.
  Control group 2: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Prime&Bond Active; Dentsply Sirona) on wet dentin in the etch-and-rinse application strategy.
  Experimental group 1: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Ambar Universal APS Plus; FGM) on overwet dentin in the etch-and-rinse application strategy.
  Experimental group 2: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Prime&Bond Active; Dentsply Sirona) on overwet dentin in the etch-and-rinse application strategy
Who Masked: Participant, Outcomes Assessor
Masking Description: Two blinded, experienced, and calibrated dentists (who specialized in esthetic dentistry with more than 15 years of clinical practice), will perform the clinical evaluation. Patients will be also blinded to group assignment. An inter-examiner and inter-examiner agreement of at least 85% will be necessary before beginning the evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): 50 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Procedure: Dentin Overwet; Device: Ambar Universal APS Plus; FGM
- Experimental group 2 (Experimental): 50 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Procedure: Dentin Overwet; Device: Prime&Bond Active; Dentsply Sirona
- Control group 1 (Active Comparator): 50 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Procedure: Dentin Wet; Device: Ambar Universal APS Plus; FGM
- Control group 2 (Active Comparator): 50 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Procedure: Dentin Wet; Device: Prime&Bond Active; Dentsply Sirona

INTERVENTIONS:
Procedure: Dentin Wet — Composite resin restorations of non-carious cervical lesions will be performed with an adhesive on wet dentin in the etch-and-rinse application strategy.
  Arms: Control group 1; Control group 2
Procedure: Dentin Overwet — Composite resin restorations of non-carious cervical lesions will be performed with an adhesive on overwet dentin in the etch-and-rinse application strategy.
  Arms: Experimental group 1; Experimental group 2
Device: Ambar Universal APS Plus; FGM — Composite resin restorations of non-carious cervical lesions will be performed with an universal adhesive
  Arms: Control group 1; Experimental group 1
Device: Prime&Bond Active; Dentsply Sirona — Composite resin restorations of non-carious cervical lesions will be performed with an universal adhesive
  Arms: Control group 2; Experimental group 2

SUMMARY:
The aim of this study will be to evaluate the effect of wet and overwet dentin on the long-term clinical performance of two universal adhesive systems used as etch-and-rinse application mode in non-carious cervical lesions (NCCLs).

Materials & Methods: 200 restorations will be randomly placed in 50 subjects according to the following groups (n=50): AMP-wet (Ambar Universal APS Plus adhesive on wet dentin); AMP-overwet (Ambar Universal APS Plus adhesive on oversaturated dentin); PBA-wet (Prime&Bond Active adhesive on wet dentin); PBA-overwet (Prime&Bond Active adhesive on oversaturated dentin). For all groups, the enamel and dentin will be etched for 15s. All groups will be light-cured for 10s/1,000 mW/cm2. A resin composite will be placed by applying three increments and each one was light cured for 20s/1,000 mW/cm2. The restorations will be finished immediately with fine diamond burs and spiral polishers. The restorations will be evaluated at baseline and after 6 months by using the FDI criteria. The following outcomes will be evaluated: retention, marginal staining, marginal adaptation, post-operative sensitivity and recurrence of caries. The differences among the groups will be calculated using Friedman repeated measures analysis of variance rank (α = 0.05).

DETAILED DESCRIPTION:
This is a four-arm, double-blind, randomized controlled clinical trial.

Control group 1: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Ambar Universal APS Plus; FGM) on wet dentin in the etch-and-rinse application strategy.

Control group 2: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Prime&Bond Active; Dentsply Sirona) on wet dentin in the etch-and-rinse application strategy.

Experimental group 1: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Ambar Universal APS Plus; FGM) on overwet dentin in the etch-and-rinse application strategy.

Experimental group 2: 50 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Prime&Bond Active; Dentsply Sirona) on overwet dentin in the etch-and-rinse application strategy

LCNCs will be randomized to universal adhesive usage and dentinal moisture levels. All groups will be light-cured with a lightcuring device (Quazar, FGM) with a light intensity of 900 mW/cm² for 10 seconds. Operators will restore the cervical area by applying three increments of resin (Llis-FGM for experimental groups 1 and 2; and TPH Spectrum-Dentsply for experimental groups 3 and 4). Each increment will light cure for 20 s at 900 mW/cm2 (Quazar, FGM). Restorations will be finished immediately with fine and extra fine diamond burs and polished with polishing spirals.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Presence of at least two Non-Carious Cervical Lesions in the dental arch with a need for restorative treatment.
* Acceptable level of oral hygiene according to the Simplified Oral Hygiene Index.
* At least 20 teeth in function.

Exclusion Criteria:

* Driving difficulties that prevent adequate oral hygiene.
* Periodontal disease.
* Active caries lesions on the teeth included in the research.
* Parafunctional habits.
* Active staples of removable partial dentures on the teeth included in the research and that these are not pillars of prostheses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Retention of restorations | From date of randomization until thirty-six four months
  Retention measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Restoration retained, no fractures / cracks;
  * G: Clinically good - Small hairline crack;
  * SS: Clinically sufficient/satisfactory - Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity);
  * US: Clinically unsatisfactory - Chipping fractures which damage marginal quality; bulk fractures with or without partial loss (less than half of the restoration);
  * PO: Clinically poor - (Partial or complete) loss of restoration, (replacement necessary).

SECONDARY OUTCOMES:
Marginal Adaptation of restorations | From date of randomization until thirty six months
  Marginal Adaptation measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Harmonious outline, no gaps, no discoloration;
  * G: Clinically good - Small marginal fracture removable by polishing;
  * SS: Clinically sufficient/satisfactory - Several small enamel or dentin fractures;
  * US: Clinically unsatisfactory - Notable enamel or dentine wall fracture;
  * PO: Clinically poor - Filling is loose but in situ.
Marginal Staining of restorations | From date of randomization until thirty six months
  Marginal Staining measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - No marginal staining;
  * G: Clinically good - Minor marginal staining, easily removable by polishing;
  * SS: Clinically sufficient/satisfactory - Moderate marginal staining, not esthetically unacceptable;
  * US: Clinically unsatisfactory - Pronounced marginal staining; major intervention necessary for improvement;
  * PO: Clinically poor - Deep marginal staining not accessible for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mario Gutierrez, PhD, Study Director — Universidad de los Andes, Chile
Locations (1):
- Mario Felipe Gutiérrez Reyes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No